CLINICAL TRIAL: NCT01597739
Title: A Phase 2a, Randomized, Multicenter, Double-blind, Placebo-controlled, Parallel-group Study of JNJ-40346527 in Subjects With Active Rheumatoid Arthritis Despite Disease-modifying Antirheumatic Drug Therapy
Brief Title: A Study of JNJ-40346527 in Patients With Active Rheumatoid Arthritis Despite Disease-modifying Antirheumatic Drug Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100801; 40346527ARA2001 (Other: Janssen Research & Development, LLC); 2011-004529-28 (EudraCT Number)
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: Active rheumatoid arthritis despite disease-modifying antirheumatic drug therapy; Disease-modifying antirheumatic drugs
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — JNJ-40346527

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JNJ-40346527 (Experimental)
  Interventions: Drug: JNJ-40346527
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-40346527 — Type=exact number; unit=mg; number=100, form=capsule; route=oral use; twice daily.
  Arms: JNJ-40346527
Drug: Placebo — Form=capsule; route=oral use; twice daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of JNJ-40346527 200 mg/day (100 mg twice daily) for 12 weeks, compared with placebo, in patients with active rheumatoid arthritis (RA) despite disease-modifying antirheumatic drug (DMARD) therapy.

DETAILED DESCRIPTION:
This is a randomized (treatment assigned by chance, like flipping a coin), multicenter, double-blind (neither physician nor patient will know the treatment the patient receives), parallel-group (each group of patients will be treated at the same time) study. JNJ-40346527 will be compared to a placebo, which is an inactive substance used to test whether a drug has a real effect. Patients will receive study medication for 12 weeks and will continue their permitted, stable DMARD therapy (methotrexate [MTX], sulfasalazine [SSZ], and/or hydroxychloroquine [HCQ]) through Week 12. A follow-up visit will occur 4 weeks after dosing is complete. The maximum length of patient participation will be 22 weeks, including a 6-week screening period. Other study visits will occur during the study, and patient safety will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (RA) for at least 6 months prior to screening
* Have been positive for, or are positive at screening for, either anti-cyclic citrullinated peptide (anti-CCP) antibody or rheumatoid factor (RF) in serum
* Have active RA with at least 6 swollen and 6 tender joints, using a 66/68 joint count at the time of screening and at baseline, and serum C-reactive protein (CRP) >= 0.80 mg/dL at screening
* Have been treated with and tolerated at least one of the following medications for a minimum of 6 months prior to screening and must be on a stable dose for a minimum of 8 weeks prior to screening: methotrexate (MTX) treatment at dosages of 7.5 to 25 mg/week, inclusive; sulfasalazine not exceeding 3 g/d; hydroxychloroquine not exceeding 400 mg/d
* If using nonsteroidal antiinflammatory drugs (NSAIDs), or other analgesics regularly for RA, patients must have been on a stable dose for at least 2 weeks prior to the first administration of study agent. If not using NSAIDs or other analgesics for RA, the patient must have not received NSAIDs or other analgesics for at least 2 weeks prior to the first administration of study agent
* If using oral corticosteroids, must be on a stable dose of <= 10 mg/day of prednisone or an equipotent dose of another oral corticosteroid for at least 2 weeks prior to the first administration of study agent. If not using corticosteroids, the patient must have not received oral corticosteroids for at least 2 weeks prior to the first administration of study agent

Exclusion Criteria:

* Has inflammatory diseases other than RA, including but not limited to adult onset Still's disease, psoriatic arthritis, ankylosing spondylitis, systemic lupus erythematosus, and Lyme disease that might confound the evaluation of the benefit of study agent therapy
* Has a history of juvenile idiopathic arthritis (JIA)
* Has current signs or symptoms of liver or renal insufficiency or cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, psychiatric, or metabolic disturbances that are severe, progressive, or uncontrolled
* Has been treated in the time frames specified with any nonbiologic disease-modifying antirheumatic drugs (DMARDs), except for MTX, sulfasazine, and hydroxychloroquine, including, but not limited to: D-penicillamine, oral or parenteral gold salts, azathioprine, cyclosporine, tacrolimus, and mycophenolate mofetil within 4 weeks prior to the first administration of study agent; leflunomide within 12 weeks prior to the first administration of study agent unless the subject has undergone a drug elimination procedure at least 4 weeks prior to the first administration of study agent; any investigational nonbiologic DMARD within 4 weeks prior to the first administration of study agent or 5 half-lives of the DMARD, whichever is longer
* Has ever received any approved or investigational biologic antirheumatic agent. These agents include, but are not limited to, infliximab, golimumab, certolizumab pegol, etanercept, adalimumab, abatacept, rituximab, tocilizumab, or anakinra.
* Has received drugs that potently inhibit or induce cytochrome P450 (CYP450) 3A4, CYP2C8, or CYP2C19 isoforms within 2 weeks or within 5 half-lives of the drug, whichever is longer, prior to the first dose of study medication
* Has received intra-articular, epidural, intravertebral, intramuscular, or intravenous corticosteroids, including adrenocorticotropic hormone, within 4 weeks prior to the first dose of study medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2012-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Disease Activity Score (DAS28), using C-reactive protein (CRP) | Week 12
  The DAS28 is a statistically derived index combining tender joints (28 joints), swollen joints (28 joints), CRP, and an overall assessment of disease activity.

SECONDARY OUTCOMES:
ACR 20 response | Week 12
  ACR 20 (American College of Rheumatology) response is a 20% improvement in rheumatoid arthritis (RA) symptoms.
DAS28 (using CRP) response | Week 12
  DAS28 response is the improvement from baseline and is rated as "No response," Moderate response," or "Good response."

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (32):
- Argentina (3):
  - Buenos Aires
  - San Juan
  - San Miguel de Tucumán
- Bulgaria (3):
  - Plovdiv
  - Sevlievo
  - Veliko Tarnovo
- Chile (2):
  - Providencia
  - Santiago
- Czechia (2):
  - Prague
  - Slaný
- Hungary (3):
  - Budapest
  - Hatvan
  - Szikszó
- Poland (3):
  - Elblag
  - Poznan
  - Warsaw
- Russia (7):
  - Kazan'
  - Moscow
  - Novosibirsk
  - Petrozavodsk
  - Saint Petersburg
  - Ulyanovsk
  - Yaroslavl
- Singapore, Singapore
- South Korea (3):
  - Gwangju
  - Seoul
  - Suwon
- Ukraine (5):
  - Donetsk
  - Kharkiv
  - Ternopil
  - Vinnitsa
  - Zaporizhzhya

REFERENCES:
- [Derived] Genovese MC, Hsia E, Belkowski SM, Chien C, Masterson T, Thurmond RL, Manthey CL, Yan XD, Ge T, Franks C, Greenspan A. Results from a Phase IIA Parallel Group Study of JNJ-40346527, an Oral CSF-1R Inhibitor, in Patients with Active Rheumatoid Arthritis despite Disease-modifying Antirheumatic Drug Therapy. J Rheumatol. 2015 Oct;42(10):1752-60. doi: 10.3899/jrheum.141580. Epub 2015 Aug 1. PMID 26233509
- See also: A Phase 2a, Randomized, Multicenter, Double-blind, Placebo-controlled, Parallel Group Study of JNJ-40346527 in Subjects With Active Rheumatoid Arthritis Despite Disease Modifying Antirheumatic Drug Therapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3469&filename=CR100801_CSR.pdf